CLINICAL TRIAL: NCT01280279
Title: Short-term Effects of Systematized Behavioral Modification Program (SBMP) for Nocturia: A Prospective Study
Brief Title: Necessity for Repetitive Education of Behavioral Modification
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Other Study IDs: nocturiaact; nocturiabehavior
Record Dates: First submitted 2011-01-17; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Patients Who Had the Urine Volume at Nighttime More Than One Third of Total Daily Urine Volume (NPU) and Voided More Than Two Times at Nighttime (Nocturia)
Keywords: Behavior modification, Behavior therapy, Nocturia, Polyuria, Quality of life
MeSH Terms: conditions — Nocturia; Polyuria | interventions — Educational Status; Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- group with nocturnal polyuria and nocturia: Patients were enrolled when they had the urine volume at nighttime more than one third of total daily urine volume (NPU) and voided more than two times at nighttime (nocturia)
  Interventions: Other: education for behavioral modification

INTERVENTIONS:
Other: education for behavioral modification — a systematized 30-minutes education program for behavioral modification (SBMP) by watching videos and discussion with a specialized continence nurse practitioner.

SUMMARY:
Few studies have reported the efficacy of repetitive education for behavioral modification as the first-line therapy for patients with nocturnal polyuria (NPU). The aim of this study is to investigate the efficacy of repetitive education for behavioral modification as the first-line therapy in the patients with NPU and to show whether a single education for behavioral modification is sufficient for the patients.

DETAILED DESCRIPTION:
Even though behavioral modification therapy seems to be effective, it is not usually recommended for patients with nocturia because much patience and understanding is required for the patients to follow the therapy. Few studies have reported the efficacy of repetitive education for behavioral modification as the first-line therapy for patients with nocturia and nocturnal polyuria (NPU). Furthermore, no report demonstrated the evidence about how many times or how long the education for behavioral therapy should be performed and how long will the education effect would continue. The aim of this study is to investigate the efficacy of repetitive education for behavioral modification as the first-line therapy in the patients with NPU and to show whether a single education for behavioral modification is sufficient for the patients.

ELIGIBILITY:
Inclusion Criteria:

* the urine volume at nighttime more than one third of total daily urine volume
* voided more than two times at nighttime

Exclusion Criteria:

* postvoid urine volume more than 100 ml
* sleep disturbance including sleep apnea
* diabetes mellitus
* diabetes insipidus
* neurogenic bladder
* congestive heart failure
* indwelling catheters
* urinary tract infection or urinary stones

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had the urine volume at nighttime more than one third of total daily urine volume (NPU) and voided more than two times at nighttime (nocturia)
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
decrease of nocturnal urine volume | 1 month after education
  The variables of FVC were prospectively collected at the time of the first visit using frequency-volume chart (FVC) for 2 days. On their second visit two weeks later, if they had nocturnal polyuria, they received the first education for behavioral modification and to fill up FVC again. When they had no improvement of nocturnal polyuria on the third visit one month later, they finally received the second education and they were recommended to fill up the FVC.

SECONDARY OUTCOMES:
improvement of symptoms and quality of life | 1 month after education
  The variables of FVC were prospectively collected at the time of the first visit using frequency-volume chart (FVC) for 2 days. On their second visit two weeks later, if they had nocturnal polyuria, they received the first education for behavioral modification and to fill up questionnaires again. When they had no improvement of nocturnal polyuria on the third visit one month later, they finally received the second education and they were recommended to fill up the FVC and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Cho, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea